CLINICAL TRIAL: NCT05153356
Title: A Prospective Longitudinal Assessment of Parkinson's Disease Functional Impairment and Disability Via Mobile Health Technology
Brief Title: A Prospective Longitudinal Assessment of PD Functional Impairment and Disability Via Mobile Health Technology
Status: Withdrawn | Type: Observational
Why Stopped: The P.I decided not to move forward with the study
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20100709
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Parkinson Disease patients: To examine the relationship between in-home continuous measures of tremor, bradykinesia, mobility, and dyskinesia acquired over a 7-day period, from 2 mobile health technologies (Personal Kinetigraph, Kinesia 360) with one-time in-clinic measures of motor functional ability pertaining to the same 7-day period as assessed by Part 2 of the MDS-UPDRS, Part 4 of the MDS-UPDRS, Neuro-QOL, and PDQ-39. This will be examined in n=20 patients (10 patients assigned to each technology with a crossover at 3 months for a total of 20 patients over 6 months, 6 timepoints with data collected every 2 weeks). Patients will then be following for an observational period of an additional 6 months.
  Interventions: Device: Personal Kinetigraph, Kinesia 360

INTERVENTIONS:
Device: Personal Kinetigraph, Kinesia 360 — 10 patients will be assigned to each technology with a crossover at 3 months for a total of 20 patients over 6 months, 6 timepoints with data collected every 2 weeks.

SUMMARY:
The purpose of this study is to compare data from a battery of novel mobile health technologies to standard-of-care validated patient questionnaires and clinician rating scales in Parkinson's disease patients.

DETAILED DESCRIPTION:
Mobile health technologies include the wearable sensor technologies that are body-worn and passively collect information and mobile devices like smartphones that can be frequently used by patients to actively or passively collect information. However, there has been limited comparison of different wearable technologies to validated clinical rating scales to allow us to come to a consensus about their utility in both clinical practice and research trials. Data from mobile health technologies in Parkinson's Disease (PD) have not been validated to use in the place of clinician rating scales. It is also not clear if the information obtained with the devices consistently correlates with change on the clinician scales and longitudinal motor decline. Technological challenges, such as the feasibility (safety, compliance) of use devices in patients with neurodegenerative disease, change in equipment and algorithms over time, collaboration with companies who may own patents, and other issues may also limit their use in healthcare and research. The purpose of this study is to compare data from a battery of novel mobile health technologies to standard-of-care validated patient questionnaires and clinician rating scales in PD patients. The hypothesis is that there will be an association between data from mobile health technologies and data obtained from validated questionnaires/scales, indicating that these technologies are a reliable means of monitoring motor symptomatology and functional impairment and disability over time. The primary aims of the study are to compare information on continuously-measured patient-reported PD-related functional impairment and disability changes from traditional validated questionnaires to continuously-measured health-related data from a battery of novel mobile health technologies, and to assess the feasibility (compliance, safety, satisfaction) of PD patients to use a battery of novel mobile health technologies.

ELIGIBILITY:
Inclusion Criteria:

* PD as defined by the UK Brain Bank Criteria
* Disease duration between 2-13 years
* Aged 35-68 years
* Hoehn & Yahr stage 3 or less when in the levodopa-"ON" state

Exclusion Criteria:

* Atypical parkinsonism including 18F-dopa PET patterns consistent with this
* MMSE score of < 24 or evidence for dementia using DSM-IV criteria
* Unable to do normal copying of interlocking pentagons and semantic fluency score <20 over 90 secs
* Ongoing major medical or psychiatric disorder including depression and psychosis
* Other concomitant treatment with neuroleptics
* Significant drug induced dyskinesias (>2 for any body part on the AIMS scale)
* Previous neurosurgery Unable to be imaged using MRI

Ages: 35 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with Parkinson Disease who are currently on levodopa treatment will be included in the study cohort. They must meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Personal Kinetigraph | 3 months
  Watch containing accelerometer and gyroscope for measurement of motor symptoms of PD
Kinesia 360 | 3 months
  2 sensor straps to wrist and ankle containing accelerometer and gyroscope for measurement of motor symptoms of PD.
MDS-UPDRS | 6 months
  Part I assesses the non-motor aspects of experiences of daily living in the week prior to the visit. Part II assesses the motor aspects of experiences of daily living in the week prior to the visit. Part III assesses motor disabilities of a subject at the time of the visit and Part IV assesses motor complications in the week prior to the visit. A total of 46 items are included in Parts I, II and III. Each item will receive a score ranging from 0 to 4 where 0 represents the absence of impairment and 4 represents the highest degree of impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Hall, MD,PhD, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.